CLINICAL TRIAL: NCT01118429
Title: Use of Oxybutynin to Treat Axillary Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo de Cirurgia Vascular (Other)
Responsible Party: Nelson Wolosker, HCFMUSP
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0083/10
Record Dates: First submitted 2010-04-29; First posted 2010-05-06 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-03

CONDITIONS: Axillary Hyperhidrosis; Osmidrosis
Keywords: hyperhidrosis; axillary; osmidrosis; oxybutynin
MeSH Terms: conditions — Body Odor; Hyperhidrosis | interventions — oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxybutynin (Experimental): Oxybutynin was prescribed for 12 weeks, in progressively increasing doses throughout treatment. At their first visit, the patients were given 2.5 mg of oxybutynin into be taken once a day in the evening, were instructed to increase the dose to 2.5 mg twice a day from the eighth to the 42nd day, and to contact the doctor if they experienced any side effect. After this period they were seen in a second visit, and the dose was increased to 5 mg twice a day from the 43rd to the end of the 84thday, to when a third visit was scheduled.
  Interventions: Drug: Oxybutynin
- Placebo (Placebo Comparator): Oxybutyinine was prescribed for 12 weeks, in progressively increasing doses throughout treatment. At their first visit, the patients were given 2.5 mg of oxybutyn into be taken once a day in the evening, were instructed to increase the dose to 2.5 mg twice a day from the eighth to the 42nd day, and to contact the doctor if they experienced any side effect. After this period they were seen in a second visit, and the dose was increased to 5 mg twice a day from the 43rd to the end of the 84thday, to when a third visit was scheduled.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxybutynin — Oxybutynin was prescribed for 12 weeks, in progressively increasing doses throughout treatment. At their first visit, the patients were given 2.5 mg of oxybutynin into be taken once a day in the evening, were instructed to increase the dose to 2.5 mg twice a day from the eighth to the 42nd day, and to contact the doctor if they experienced any side effect. After this period they were seen in a second visit, and the dose was increased to 5 mg twice a day from the 43rd to the end of the 84thday, to when a third visit was scheduled.
  Arms: Oxybutynin
Drug: Placebo — Oxybutyinine was prescribed for 12 weeks, in progressively increasing doses throughout treatment. At their first visit, the patients were given 2.5 mg of oxybutyn into be taken once a day in the evening, were instructed to increase the dose to 2.5 mg twice a day from the eighth to the 42nd day, and to contact the doctor if they experienced any side effect. After this period they were seen in a second visit, and the dose was increased to 5 mg twice a day from the 43rd to the end of the 84thday, to when a third visit was scheduled.
  Arms: Placebo

SUMMARY:
The objective of this study was to evaluate the effectiveness and patient satisfaction with the use of oxybutynin at low doses for treating axillary hyperhidrosis in a large series of patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with axillary hyperhidrosis

Exclusion Criteria:

* glaucoma and micturition disorders, pregnancy

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of treatment by a clinical questionnaire | 6 weeks of treatment
  These evaluations were used to assess (1) the patients' clinical improvement in axillary hyperhidrosis, using a clinical questionnaire, published at 2003:
  de Campos JR, Kauffman P, Werebe Ede C, Andrade Filho LO, Kusniek S, Wolosker N, Jatene FB.Quality of life, before and after thoracic sympathectomy: report on 378 operated patients.Ann Thorac Surg. 2003 Sep;76(3):886-91
Effectiveness of treatment using a clinical questionnaire | After 12 weeks of treatment
  These evaluations were used to assess (1) the patients' clinical improvement in axillary hyperhidrosis, using a clinical questionnaire:
  de Campos JR, Kauffman P, Werebe Ede C, Andrade Filho LO, Kusniek S, Wolosker N, Jatene FB.Quality of life, before and after thoracic sympathectomy: report on 378 operated patients.Ann Thorac Surg. 2003 Sep;76(3):886-91

SECONDARY OUTCOMES:
Treatment of hyperhidrosis at other sites | 6 weeks
  These evaluations were used to assess (1) the patients' clinical improvement in hyperhidrosis at other sites, using a clinical questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Wolosker, MD, PhD, Principal Investigator — Hospital das Clinicas, University of Sao Paulo
Locations (1):
- Hospital das Clinicas da FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Wolosker N, Yazbek G, de Campos JR, Munia MA, Kauffman P, Jatene FB, Puech-Leao P. Quality of life before surgery is a predictive factor for satisfaction among patients undergoing sympathectomy to treat hyperhidrosis. J Vasc Surg. 2010 May;51(5):1190-4. doi: 10.1016/j.jvs.2009.11.078. Epub 2010 Mar 29. PMID 20299178
- [Background] de Campos JR, Wolosker N, Yazbek G, Munia MA, Kauffman P, Puech-Leao P, Jatene FB. Comparison of pain severity following video-assisted thoracoscopic sympathectomy: electric versus harmonic scalpels. Interact Cardiovasc Thorac Surg. 2010 Jun;10(6):919-22. doi: 10.1510/icvts.2009.225383. Epub 2010 Mar 16. PMID 20233806
- [Background] Yazbek G, Wolosker N, Kauffman P, Campos JR, Puech-Leao P, Jatene FB. Twenty months of evolution following sympathectomy on patients with palmar hyperhidrosis: sympathectomy at the T3 level is better than at the T2 level. Clinics (Sao Paulo). 2009;64(8):743-9. doi: 10.1590/S1807-59322009000800006. PMID 19690657
- [Background] Munia MA, Wolosker N, Kaufmann P, de Campos JR, Puech-Leao P. Sustained benefit lasting one year from T4 instead of T3-T4 sympathectomy for isolated axillary hyperhidrosis. Clinics (Sao Paulo). 2008 Dec;63(6):771-4. doi: 10.1590/s1807-59322008000600011. PMID 19060999
- [Background] Wolosker N, Yazbek G, Ishy A, de Campos JR, Kauffman P, Puech-Leao P. Is sympathectomy at T4 level better than at T3 level for treating palmar hyperhidrosis? J Laparoendosc Adv Surg Tech A. 2008 Feb;18(1):102-6. doi: 10.1089/lap.2007.0030. PMID 18266585
- [Background] Munia MA, Wolosker N, Kauffman P, de Campos JR, Puech-Leao P. A randomized trial of T3-T4 versus T4 sympathectomy for isolated axillary hyperhidrosis. J Vasc Surg. 2007 Jan;45(1):130-3. doi: 10.1016/j.jvs.2006.09.011. PMID 17210397